CLINICAL TRIAL: NCT01664910
Title: Anti-CD22 Immunoconjugate Inotuzumab Ozogamicin (CMC-544) Added to Fludarabine, Bendamustine and Rituximab and Allogeneic Transplantation for CD22 Positive-Lymphoid Malignancies
Brief Title: CMC-544 and Allogeneic Transplantation for CD22 Positive-Lymphoid Malignancies
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2012-0265; NCI-2012-02072 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2012-0265 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2012-08-10; First posted 2012-08-14 (Estimated); Results first posted 2024-07-23 (Actual); Last update posted 2024-07-23 (Actual); Status verified 2024-06

CONDITIONS: Hematopoietic and Lymphoid Cell Neoplasm
MeSH Terms: conditions — Hematologic Neoplasms | interventions — Antilymphocyte Serum; thymoglobulin; Bendamustine Hydrochloride; fludarabine phosphate; Inotuzumab Ozogamicin; Methotrexate; merphos; Peripheral Blood Stem Cell Transplantation; Rituximab; CT-P10; Tacrolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (transplant) (Experimental): Patients receive inotuzumab ozogamicin IV over 1 hour on day -13, and fludarabine phosphate IV over 1 hour and bendamustine hydrochloride IV over 30 minutes to 1 hour on days -5 to -3. Patients with CD20-positive disease also receive rituximab IV over 4-6 hours on days -6, 1, and 8 and patients with MUD receive anti-thymocyte globulin IV over 3-4 hours on days -2 to -1. All patients also receive tacrolimus IV over 24 hours continuously or PO daily beginning on days -2 to 180 followed by taper in the absence of GVHD and methotrexate IV over 30 minutes on days 1, 3, and 6 (1, 3, 6, and 11 in patients with MUD). Patients undergo allogeneic BM or PBSC transplant on day 0.
  Interventions: Procedure: Allogeneic Bone Marrow Transplantation; Procedure: Allogeneic Hematopoietic Stem Cell Transplantation; Biological: Anti-Thymocyte Globulin; Drug: Bendamustine Hydrochloride; Drug: Fludarabine Phosphate; Biological: Inotuzumab Ozogamicin; Drug: Methotrexate; Procedure: Peripheral Blood Stem Cell Transplantation; Biological: Rituximab; Drug: Tacrolimus

INTERVENTIONS:
Procedure: Allogeneic Bone Marrow Transplantation — Undergo allogeneic BM transplant
  Other Names: Allo BMT; Allogeneic BMT
Procedure: Allogeneic Hematopoietic Stem Cell Transplantation — Undergo allogeneic PBSC or BM transplant
  Other Names: Allogeneic Hematopoietic Cell Transplantation; Allogeneic Stem Cell Transplantation; HSC; HSCT
Biological: Anti-Thymocyte Globulin — Given IV
  Other Names: Antithymocyte Globulin; Antithymocyte Serum; ATG; ATGAM; ATS; Thymoglobulin
Drug: Bendamustine Hydrochloride — Given IV
  Other Names: Bendamustin Hydrochloride; Cytostasan Hydrochloride; Levact; Ribomustin; SyB L-0501; Treanda
Drug: Fludarabine Phosphate — Given IV
  Other Names: 2-F-ara-AMP; 9H-Purin-6-amine, 2-fluoro-9-(5-O-phosphono-.beta.-D-arabinofuranosyl)-; Beneflur; Fludara; SH T 586
Biological: Inotuzumab Ozogamicin — Given IV
  Other Names: Besponsa; CMC-544; Way 207294; WAY-207294
Drug: Methotrexate — Given IV
  Other Names: Abitrexate; Alpha-Methopterin; Amethopterin; Brimexate; CL 14377; CL-14377; Emtexate; Emthexat; Emthexate; Farmitrexat; Fauldexato; Folex; Folex PFS; Lantarel; Ledertrexate; Lumexon; Maxtrex; Medsatrexate; Metex; Methoblastin; Methotrexate LPF; Methotrexate Methylaminopterin; Methotrexatum; Metotrexato; Metrotex; Mexate; Mexate-AQ; MTX; Novatrex; Rheumatrex; Texate; Tremetex; Trexeron; Trixilem; WR-19039
Procedure: Peripheral Blood Stem Cell Transplantation — Undergo allogeneic PBSC transplant
  Other Names: PBPC transplantation; PBSCT; Peripheral Blood Progenitor Cell Transplantation; Peripheral Stem Cell Support; Peripheral Stem Cell Transplant; Peripheral Stem Cell Transplantation
Biological: Rituximab — Given IV
  Other Names: ABP 798; BI 695500; C2B8 Monoclonal Antibody; Chimeric Anti-CD20 Antibody; CT-P10; IDEC-102; IDEC-C2B8; IDEC-C2B8 Monoclonal Antibody; MabThera; Monoclonal Antibody IDEC-C2B8; PF-05280586; Rituxan; Rituximab Biosimilar ABP 798; Rituximab Biosimilar BI 695500; Rituximab Biosimilar CT-P10; Rituximab Biosimilar GB241; Rituximab Biosimilar IBI301; Rituximab Biosimilar PF-05280586; Rituximab Biosimilar RTXM83; Rituximab Biosimilar SAIT101; RTXM83
Drug: Tacrolimus — Given IV or PO
  Other Names: FK 506; Fujimycin; Hecoria; Prograf; Protopic

SUMMARY:
This phase I/II trial studies the side effects and the best dose of inotuzumab ozogamicin when given together with fludarabine phosphate, bendamustine hydrochloride, and rituximab before donor stem cell transplant in treating patients with lymphoid malignancies. Giving chemotherapy drugs, such as fludarabine phosphate and bendamustine hydrochloride, before a donor peripheral blood stem cell transplant helps stop the growth of cancer cells or abnormal cell and helps stop the patient's immune system from rejecting the donor's stem cells. Immunotherapy with monoclonal antibodies, such as inotuzumab ozogamicin and rituximab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. When the healthy stem cells from a donor are infused into the patient they may help the patient's bone marrow make stem cells, red blood cells, white blood cells, and platelets. Sometimes the transplanted cell from a donor can make an immune system response against the body's normal cells. Giving fludarabine phosphate and bendamustine hydrochloride before the transplant together with anti-thymocyte globulin and tacrolimus may stop this from happening.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To characterize the safety of anti-cluster of differentiation (CD) 22 immunoconjugate inotuzumab ozogamicin (CMC-544), when administered in conjunction with fludarabine (fludarabine phosphate), bendamustine (bendamustine hydrochloride), and rituximab as non-myeloablative preparative regimen for allogeneic stem cell transplantation for CD22-positive lymphoid malignancies.

SECONDARY OBJECTIVES:

I. To estimate tumor response. II. To determine overall and event-free survival rates by histology subtype.

OUTLINE: This is a dose-escalation study of inotuzumab ozogamicin.

Patients receive inotuzumab ozogamicin intravenously (IV) over 1 hour on day -13, and fludarabine phosphate IV over 1 hour and bendamustine hydrochloride IV over 30 minutes to 1 hour on days -5 to -3. Patients with CD20-positive disease also receive rituximab IV over 4-6 hours on days -6, 1, and 8 and patients with matched unrelated donors (MUD) receive anti-thymocyte globulin IV over 3-4 hours on days -2 to -1. All patients also receive tacrolimus IV over 24 hours continuously or orally (PO) daily beginning on days -2 to 180 followed by taper in the absence of graft-versus-host disease (GVHD) and methotrexate IV over 30 minutes on days 1, 3, and 6 (1, 3, 6, and 11 in patients with MUD). Patients undergo allogeneic bone marrow (BM) or peripheral blood stem cell (PBSC) transplant on day 0.

After completion of study treatment, patients are followed up periodically.

ELIGIBILITY:
Inclusion Criteria:

* Patients with B-cell hematological malignancies who are eligible for allogeneic transplantation
* Patients must have a fully-matched sibling donor or a matched unrelated donor identified
* Performance score of at least 80% by Karnofsky or 0 to 2 Eastern Cooperative Oncology Group (ECOG)
* Left ventricular ejection fraction (EF) >= 45% with no uncontrolled arrhythmias or symptomatic heart disease
* Forced expiratory volume in one second (FEV1) >= 50%
* Forced vital capacity (FVC) >= 50%
* Corrected diffusion capacity of the lung for carbon monoxide (DLCO) >= 50%
* Serum creatinine < 1.6 mg/dL
* Serum bilirubin < 2 mg/dL upper limit of normal (unless due to Gilbert's disease; patient with this disease should have a right upper quadrant ultrasound evaluation before treatment)
* Serum glutamate pyruvate transaminase (SGPT) < 2 x upper limit of normal
* Men and women of reproductive potential must agree to follow accepted birth control methods (i.e., a hormonal contraceptive, intra-uterine device, diaphragm with spermicide, condom with spermicide, or abstinence) for the duration of the study
* Negative beta human chorionic gonadotropin (HCG) test in a woman with child bearing potential (defined as not post-menopausal for 12 months or no previous surgical sterilization) or currently breast-feeding; pregnancy testing is not required for post-menopausal or surgically sterilized women

Exclusion Criteria:

* Patient with active central nervous system (CNS) involvement
* Known infection with human immunodeficiency virus (HIV), human T-cell lymphotropic virus (HTLV)-I, hepatitis B, or hepatitis C
* Patients with other malignancies diagnosed within 2 years prior to study registration; skin squamous or basal cell carcinoma are exceptions
* Active bacterial, viral or fungal infections
* History of stroke within 6 months
* History of biliary colic attack
* A prior autologous transplant within 3 months of study entry or allogeneic stem cell transplant
* Serious medical or psychiatric illness likely to interfere with participation in this clinical study
* Patient has received other investigational drugs within 3 weeks before study registration
* Serious nonmalignant disease which, in the opinion of the investigator would compromise protocol objectives
* Prior exposure to CMC-544 within past 6 months
* Established refractoriness to CMC-544

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2012-10-29 (Actual); Primary Completion 2023-06-28 (Actual); Study Completion 2023-06-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Issa Khouri, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All recruitment done at the University of Texas MD Anderson Cancer Center.
Groups:
- Cohort 1:Allogeneic TP for CD22(+) Lymphoid Malignancy Conditioned w/ Flu/Ben/Rit/CMC544(0.6 mg/m2): Patients receive inotuzumab ozogamicin IV over 1 hour on day -13, and fludarabine phosphate IV over 1 hour and bendamustine hydrochloride IV over 30 minutes to 1 hour on days -5 to -3. Patients with CD20-positive disease also receive rituximab IV over 4-6 hours on days -6, 1, and 8 and patients with MUD receive anti-thymocyte globulin IV over 3-4 hours on days -2 to -1. All patients also receive tacrolimus IV over 24 hours continuously or PO daily beginning on days -2 to 180 followed by taper in the absence of GVHD and methotrexate IV over 30 minutes on days 1, 3, and 6 (1, 3, 6, and 11 in patients with MUD). Patients undergo allogeneic BM or PBSC transplant on day 0.
  Allogeneic Bone Marrow Transplantation: Undergo allogeneic BM transplant
  Allogeneic Hematopoietic Stem Cell Transplantation: Undergo allogeneic PBSC or BM transplant
  Anti-Thymocyte Globulin: Given IV
  Bendamustine Hydrochloride: Given IV
  Fludarabine Phosphate: Given IV
  Inotuzumab Ozogamicin: Given IV at 0.6 mg/m2
  Methotrexate: Given IV
  Peripheral Blood Stem Cell Transplantation: Undergo allogeneic PBSC transplant
  Rituximab: Given IV
  Tacrolimus: Given IV or PO
- Cohort 2:Allogeneic TP for CD22(+) Lymphoid Malignancy Conditioned w/ Flu/Ben/Rit/CMC544(1.2 mg/m2): Patients receive inotuzumab ozogamicin IV over 1 hour on day -13, and fludarabine phosphate IV over 1 hour and bendamustine hydrochloride IV over 30 minutes to 1 hour on days -5 to -3. Patients with CD20-positive disease also receive rituximab IV over 4-6 hours on days -6, 1, and 8 and patients with MUD receive anti-thymocyte globulin IV over 3-4 hours on days -2 to -1. All patients also receive tacrolimus IV over 24 hours continuously or PO daily beginning on days -2 to 180 followed by taper in the absence of GVHD and methotrexate IV over 30 minutes on days 1, 3, and 6 (1, 3, 6, and 11 in patients with MUD). Patients undergo allogeneic BM or PBSC transplant on day 0.
  Allogeneic Bone Marrow Transplantation: Undergo allogeneic BM transplant
  Allogeneic Hematopoietic Stem Cell Transplantation: Undergo allogeneic PBSC or BM transplant
  Anti-Thymocyte Globulin: Given IV
  Bendamustine Hydrochloride: Given IV
  Fludarabine Phosphate: Given IV
  Inotuzumab Ozogamicin: Given IV at 1.2 mg/m2
  Methotrexate: Given IV
  Peripheral Blood Stem Cell Transplantation: Undergo allogeneic PBSC transplant
  Rituximab: Given IV
  Tacrolimus: Given IV or PO
- Cohort 3:Allogeneic TP for CD22(+) Lymphoid Malignancy Conditioned w/ Flu/Ben/Rit/CMC544(1.8 mg/m2): Patients receive inotuzumab ozogamicin IV over 1 hour on day -13, and fludarabine phosphate IV over 1 hour and bendamustine hydrochloride IV over 30 minutes to 1 hour on days -5 to -3. Patients with CD20-positive disease also receive rituximab IV over 4-6 hours on days -6, 1, and 8 and patients with MUD receive anti-thymocyte globulin IV over 3-4 hours on days -2 to -1. All patients also receive tacrolimus IV over 24 hours continuously or PO daily beginning on days -2 to 180 followed by taper in the absence of GVHD and methotrexate IV over 30 minutes on days 1, 3, and 6 (1, 3, 6, and 11 in patients with MUD). Patients undergo allogeneic BM or PBSC transplant on day 0.
  Allogeneic Bone Marrow Transplantation: Undergo allogeneic BM transplant
  Allogeneic Hematopoietic Stem Cell Transplantation: Undergo allogeneic PBSC or BM transplant
  Anti-Thymocyte Globulin: Given IV
  Bendamustine Hydrochloride: Given IV
  Fludarabine Phosphate: Given IV
  Inotuzumab Ozogamicin: Given IV at 1.8 mg/m2
  Methotrexate: Given IV
  Peripheral Blood Stem Cell Transplantation: Undergo allogeneic PBSC transplant
  Rituximab: Given IV
  Tacrolimus: Given IV or PO
Period: Overall Study
Arm/Group | Cohort 1:Allogeneic TP for CD22(+) Lymphoid Malignancy Conditioned w/ Flu/Ben/Rit/CMC544(0.6 mg/m2) | Cohort 2:Allogeneic TP for CD22(+) Lymphoid Malignancy Conditioned w/ Flu/Ben/Rit/CMC544(1.2 mg/m2) | Cohort 3:Allogeneic TP for CD22(+) Lymphoid Malignancy Conditioned w/ Flu/Ben/Rit/CMC544(1.8 mg/m2)
Started | 4 | 2 | 21
Completed | 4 | 2 | 20
Not Completed | 0 | 0 | 1
Not completed — Adverse Event | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1:Allogeneic TP for CD22(+) Lymphoid Malignancy Conditioned w/ Flu/Ben/Rit/CMC544(0.6 mg/m2) | Cohort 2:Allogeneic TP for CD22(+) Lymphoid Malignancy Conditioned w/ Flu/Ben/Rit/CMC544(1.2 mg/m2) | Cohort 3:Allogeneic TP for CD22(+) Lymphoid Malignancy Conditioned w/ Flu/Ben/Rit/CMC544(1.8 mg/m2) | Total
Number analyzed (Participants) | 4 | 2 | 21 | 27
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 4 | 2 | 17 | 23
  >=65 years | 0 | 0 | 4 | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 0 | 8 | 12
  Male | 0 | 2 | 13 | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 2 | 2
  Not Hispanic or Latino | 4 | 2 | 19 | 25
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 4 | 2 | 21 | 27

OUTCOME MEASURES:

1. Primary Outcome: Maximum-tolerated Dose (MTD) of Inotuzumab Without DLT
Description: Number of participants received inotuzumab in each cohort without DLT
Time Frame: Up to 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1:Allogeneic TP for CD22(+) Lymphoid Malignancy Conditioned w/ Flu/Ben/Rit/CMC544(0.6 mg/m2) | Cohort 2:Allogeneic TP for CD22(+) Lymphoid Malignancy Conditioned w/ Flu/Ben/Rit/CMC544(1.2 mg/m2) | Cohort 3:Allogeneic TP for CD22(+) Lymphoid Malignancy Conditioned w/ Flu/Ben/Rit/CMC544(1.8 mg/m2)
Number analyzed (Participants) | 4 | 2 | 21
Participants | 4 | 2 | 20

2. Secondary Outcome: Overall Response
Description: Overall response (CR+PR) with estimated with a 95% confidence interval in the dose that is declared the MTD. Complete Response is no clinical or radiological evidence of disease. Partial remission is equal to or more than 50% reduction in lymphadenopathy, liver and or spleen if abnormal at pre-treatment.
Time Frame: Up to 3 years
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1:Allogeneic TP for CD22(+) Lymphoid Malignancy Conditioned w/ Flu/Ben/Rit/CMC544(0.6 mg/m2) | Cohort 2:Allogeneic TP for CD22(+) Lymphoid Malignancy Conditioned w/ Flu/Ben/Rit/CMC544(1.2 mg/m2) | Cohort 3:Allogeneic TP for CD22(+) Lymphoid Malignancy Conditioned w/ Flu/Ben/Rit/CMC544(1.8 mg/m2)
Number analyzed (Participants) | 4 | 2 | 21
Participants
  Complete Response | 4 | 2 | 19
  Partial Response | 0 | 0 | 1
  Not Evaluable | 0 | 0 | 1

3. Secondary Outcome: Overall Survival (OS)
Description: Participants are disease free and alive at 3 years post transplant.
Time Frame: Up to 3 years
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1:Allogeneic TP for CD22(+) Lymphoid Malignancy Conditioned w/ Flu/Ben/Rit/CMC544(0.6 mg/m2) | Cohort 2:Allogeneic TP for CD22(+) Lymphoid Malignancy Conditioned w/ Flu/Ben/Rit/CMC544(1.2 mg/m2) | Cohort 3:Allogeneic TP for CD22(+) Lymphoid Malignancy Conditioned w/ Flu/Ben/Rit/CMC544(1.8 mg/m2)
Number analyzed (Participants) | 4 | 2 | 21
Participants | 4 | 2 | 14

ADVERSE EVENTS:
Time Frame: Up to 3 years
Arm/Group | Cohort 1:Allogeneic TP for CD22(+) Lymphoid Malignancy Conditioned w/ Flu/Ben/Rit/CMC544(0.6 mg/m2) | Cohort 2:Allogeneic TP for CD22(+) Lymphoid Malignancy Conditioned w/ Flu/Ben/Rit/CMC544(1.2 mg/m2) | Cohort 3:Allogeneic TP for CD22(+) Lymphoid Malignancy Conditioned w/ Flu/Ben/Rit/CMC544(1.8 mg/m2)
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/2 | 7/21
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/2 | 2/21
Other Adverse Events (participants affected / at risk) | 4/4 | 2/2 | 16/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1:Allogeneic TP for CD22(+) Lymphoid Malignancy Conditioned w/ Flu/Ben/Rit/CMC544(0.6 mg/m2) (N=4) | Cohort 2:Allogeneic TP for CD22(+) Lymphoid Malignancy Conditioned w/ Flu/Ben/Rit/CMC544(1.2 mg/m2) (N=2) | Cohort 3:Allogeneic TP for CD22(+) Lymphoid Malignancy Conditioned w/ Flu/Ben/Rit/CMC544(1.8 mg/m2) (N=21)
Bacterial (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
Encephalopathy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
HSCT related microangiopathy (TA-TMA) (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
DAH (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2)
GI GvHD (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2)
Chronic GI GvHD (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Liver GvHD (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1:Allogeneic TP for CD22(+) Lymphoid Malignancy Conditioned w/ Flu/Ben/Rit/CMC544(0.6 mg/m2) (N=4) | Cohort 2:Allogeneic TP for CD22(+) Lymphoid Malignancy Conditioned w/ Flu/Ben/Rit/CMC544(1.2 mg/m2) (N=2) | Cohort 3:Allogeneic TP for CD22(+) Lymphoid Malignancy Conditioned w/ Flu/Ben/Rit/CMC544(1.8 mg/m2) (N=21)
Diarrhea (Gastrointestinal disorders) | 2 (2) | 0 (0) | 4 (4)
Nausea (Gastrointestinal disorders) | 4 (4) | 1 (1) | 16 (16)
ATG fevers (General disorders) | 2 (2) | 0 (0) | 0 (0)
Fluid overload (General disorders) | 1 (1) | 0 (0) | 10 (10)
Bacterial Infection (Infections and infestations) | 2 (2) | 1 (1) | 8 (8)
Viral Infections (Infections and infestations) | 3 (3) | 1 (1) | 11 (11)
Elevated bilirubin (Investigations) | 1 (1) | 0 (0) | 3 (3)
Arthralgia due to Chronic GvHD (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
BK virus induced hemohrragic cystitis (Renal and urinary disorders) | 1 (1) | 0 (0) | 2 (2)
Chronic lung GvHD (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Chronic skin GvHD (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 9 (9)
Skin GvHD (Skin and subcutaneous tissue disorders) | 3 (3) | 1 (1) | 8 (8)
Skin rash due to ATG (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Neutropenic fevers (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 1 (1)
Chronic ocular GvHD (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Chronic oral GvHD (Gastrointestinal disorders) | 0 (0) | 2 (2) | 10 (10)
GI GvHD (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Fevers (General disorders) | 0 (0) | 1 (1) | 7 (7)
Skin rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Ascitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Chronic GI GvHD (Gastrointestinal disorders) | 0 (0) | 0 (0) | 3 (3)
Chronic GvHD_Fascitis (General disorders) | 0 (0) | 0 (0) | 5 (5)
Chronic liver GvHD (Hepatobiliary disorders) | 0 (0) | 0 (0) | 5 (5)
Chronic vaginal GvHD (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 3 (3)
Creatinine increased (Investigations) | 0 (0) | 0 (0) | 3 (3)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Ejection fraction decreased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Elevated transminitis (General disorders) | 0 (0) | 0 (0) | 3 (3)
Flu like syndrome (General disorders) | 0 (0) | 0 (0) | 1 (1)
Fungal Infections (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 3 (3)
Ocular GvHD (Eye disorders) | 0 (0) | 0 (0) | 5 (5)
Orthostatic hypotension (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 3 (3)
Venous occlusive disease (General disorders) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-11-09): https://cdn.clinicaltrials.gov/large-docs/10/NCT01664910/Prot_SAP_000.pdf